CLINICAL TRIAL: NCT00004205
Title: A Phase III Study to Evaluate Letrozole as Adjuvant Endocrine Therapy for Postmenopausal Women With Receptor (ER and/or PgR) Positive Tumors
Brief Title: Letrozole or Tamoxifen in Treating Postmenopausal Women With Breast Cancer
Acronym: BIG 1-98
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: UNICANCER (Other); Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000067451; IBCSG-18-98; DAN-DBCG-IBCSG-1-98; FRE-FNCLCC-IBCSG-1-98; EU-99022; NOVARTIS-2026703019; BIG-1-98
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; breast cancer in situ; recurrent breast cancer; ductal breast carcinoma; lobular breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Ductal, Breast | interventions — Letrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tamoxifen (Experimental): Tamoxifen for 5 years after randomization.
  Interventions: Drug: tamoxifen citrate
- Letrozole (Experimental): Letrozole for 5 years after randomization.
  Interventions: Drug: letrozole
- Tamoxifen, then letrozole (Experimental): Tamoxifen for 2 years after randomization, then letrozole for the next 3 years.
  Interventions: Drug: letrozole; Drug: tamoxifen citrate
- Letrozole, then tamoxifen (Experimental): Letrozole for 2 years after randomization, then tamoxifen for the next 3 years.
  Interventions: Drug: letrozole; Drug: tamoxifen citrate

INTERVENTIONS:
Drug: letrozole — Letrozole 2.5 mg daily oral administration.
  Arms: Letrozole; Letrozole, then tamoxifen; Tamoxifen, then letrozole
Drug: tamoxifen citrate — Tamoxifen 20 mg daily oral administration.
  Arms: Letrozole, then tamoxifen; Tamoxifen; Tamoxifen, then letrozole

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by reducing the production of estrogen. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells. If is not yet known which treatment regimen is most effective for breast cancer.

PURPOSE: Randomized double-blind phase III trial to compare the effectiveness of letrozole with that of tamoxifen in treating postmenopausal women who have breast cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare adjuvant letrozole vs tamoxifen administered for 5 years in postmenopausal women with operable, hormone receptor-positive breast cancer.
* Compare these treatment regimens given sequentially vs continuously in this patient population.
* Compare these treatment regimens in terms of overall survival, disease-free and systemic-free survival, safety, and tolerability in this patient population.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to adjuvant chemotherapy (prior therapy vs no prior or concurrent therapy vs concurrent therapy), prior surgery (modified radical mastectomy vs a lesser surgical procedure), and participating center. Patients are randomized to one of four treatment arms.

* Arm I: Patients receive adjuvant oral tamoxifen daily for 5 years.
* Arm II: Patients receive adjuvant oral letrozole daily for 5 years.
* Arm III: Patients receive adjuvant oral tamoxifen daily for 2 years followed by adjuvant oral letrozole daily for 3 years.
* Arm IV: Patients receive adjuvant oral letrozole daily for 2 years followed by adjuvant oral tamoxifen daily for 3 years.

Patients may receive concurrent radiotherapy. Some patients receive concurrent adjuvant chemotherapy beginning within 8 weeks after surgery and continuing for no more than 6 months.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 5,180 patients (1,295 per treatment arm) will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed resectable adenocarcinoma of the breast

  * pT1, pT2, pT3, or minimal dermal involvement on pathology only
  * pN0, pN1, pN2, or M0

    * Negative nodal status

      * At least 8 nodes are negative
    * Unknown nodal status

      * Less than 8 nodes examined and no pathological finding
    * Positive nodal status

      * Any positive finding independent of the number of nodes examined
  * Negative sentinel node or no prior nodal dissection allowed if all other criteria met
* Must have had total mastectomy, lumpectomy, or quadrantectomy

  * Should have prior chest wall radiotherapy after segmental mastectomy or histopathologic T4 dermal involvement
* Stage I, II, or IIIa allowed if the tumor is completely removed macroscopically and margins of the resected tumor are microscopically free of tumor
* Must undergo chest wall radiotherapy or second resection if microscopic disease at the mastectomy margins
* No bilateral disease except in situ disease, either ductal or lobular of the contralateral breast
* Postmenopausal

  * Regardless of prior hormonal replacement therapy (HRT) or hysterectomy:

    * Bilateral oophorectomy and any age
    * Radiologic castration and amenorrheic for at least 3 months and any age
    * Not postmenopausal at the start of adjuvant chemotherapy AND and completed at least 6 courses of prior cyclophosphamide, methotrexate, and fluorouracil (CMF) or at least 4 courses of prior anthracycline-cyclophosphamide continuation therapy and at least age 45 with follicle stimulating hormone (FSH), luteinizing hormone (LH), and estradiol (E2) postmenopausal levels
  * No prior HRT:

    * Prior hysterectomy and less than age 55 with FSH/LH/E2 postmenopausal levels
    * Prior hysterectomy and at least age 55
  * No prior HRT or hysterectomy:

    * Amenorrhea more than 1 year and less than age 50
    * Amenorrhea more than 6 months and at least age 50
  * Prior HRT regardless of hysterectomy:

    * At least 1 month since prior HRT and less than age 55 with FSH/LH/E2 postmenopausal levels
    * At least 1 month since prior HRT and at least age 55
  * FSH/LH/E2 postmenopausal levels and uncategorized
* No distant metastases, including bone scans showing hot spots unconfirmed as benign disease or skeletal pain of unknown cause
* At least 10% hormone receptor-positive tumor cells
* Hormone receptor status:

  * Estrogen receptor positive AND/OR
  * Progesterone receptor positive

PATIENT CHARACTERISTICS:

Age:

* 30 and over

Sex:

* Female

Menopausal status:

* Postmenopausal

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than 3.0 mg/dL
* SGOT or SGPT less than 1.5 times upper limit of normal
* No hepatic disease that would preclude study

Renal:

* Creatinine less than 1.8 mg/dL
* No renal disease that would preclude study

Cardiovascular:

* No cardiovascular disease that would preclude study
* Prior deep vein thrombosis allowed if medically stable

Pulmonary:

* No lung embolism

Other:

* No other prior or concurrent malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No prior noncompliance to medical regimens
* No other nonmalignant systemic diseases that would preclude follow-up
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior immunotherapy or biological response modifiers (e.g., interferon) allowed

Chemotherapy:

* See Disease Characteristics
* Prior adjuvant or neoadjuvant chemotherapy allowed
* Concurrent adjuvant chemotherapy allowed

Endocrine therapy:

* See Disease Characteristics
* Prior neoadjuvant hormonal therapy allowed (e.g., antiestrogens, progestins, or aromatase inhibitors) if no more than 4 months duration and no disease progression
* Prior corticosteroids allowed
* At least 4 weeks since prior HRT
* Prior adjuvant antiestrogen therapy allowed if less than 1 month duration and immediately after surgery, radiotherapy, and/or chemotherapy
* Prior antiestrogens for chemoprevention allowed if at least 18 months between completion of chemoprevention and diagnosis
* No other concurrent antiestrogens or aromatase inhibitors
* No concurrent raloxifene
* No concurrent systemic HRT with or without progestins of more than 3 months duration

Radiotherapy:

* See Disease Characteristics
* Concurrent radiotherapy allowed

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior systemic investigational drugs
* At least 7 days since prior topical investigational drugs
* Concurrent bisphosphonates allowed

Ages: 30 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8028 (Actual)
Dates: Start 1998-03; Primary Completion 2008-12 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Disease free survival. | Up to end of year 2015
  Time from randomization to recurrence (including recurrence restricted to the breast after breast conserving treatment), metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to end of year 2015, for a maximum of 17 years

SECONDARY OUTCOMES:
Overall survival | Up to end of year 2015
  Time from randomization to death from any cause, assessed up to end of year 2015, for a maximum of 17 years
Safety | 5 years after randomization.
  Morbidity information will be recorded using the Adverse Event Form (AE).
Systemic relapse | Up to end of year 2015
  Time from randomization to appearance of any recurrent or metastatic disease in sites other than the local mastectomy scar, the ipsilateral breast in case of breast conservation, or the contralateral breast, assessed up to end of year 2015, for a maximum of 17 years

CONTACTS AND LOCATIONS:
Overall Officials: Beat Thurlimann, MD, Study Chair — Cantonal Hospital of St. Gallen; Louis Mauriac, MD, Study Chair — Institut Bergonié; Henning T. Mouridsen, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (3):
- Rigshospitalet, Copenhagen, Denmark
- Institut Bergonie, Bordeaux, France
- Kantonsspital - St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Lipsitz M, Delea TE, Guo A. Cost effectiveness of letrozole versus anastrozole in postmenopausal women with HR+ early-stage breast cancer. Curr Med Res Opin. 2010 Oct;26(10):2315-28. doi: 10.1185/03007995.2010.510784. PMID 20731528
- [Background] Skedgel C, Rayson D, Younis T, et al.: Direct and indirect economic evaluation of upfront and sequential adjuvant treatment in postmenopausal women with breast cancer based on the BIG 1-98 trial. [Abstract] J Clin Oncol 27 (Suppl 15): A-6594, 2009.
- [Background] Delea TE, El-Ouagari K, Karnon J, Sofrygin O. Cost-effectiveness of letrozole versus tamoxifen as initial adjuvant therapy in postmenopausal women with hormone-receptor positive early breast cancer from a Canadian perspective. Breast Cancer Res Treat. 2008 Apr;108(3):375-87. doi: 10.1007/s10549-007-9607-7. Epub 2007 Jul 26. PMID 17653859
- [Background] Delea TE, Karnon J, Sofrygin O, Thomas SK, Papo NL, Barghout V. Cost-effectiveness of letrozole versus tamoxifen as initial adjuvant therapy in hormone receptor-positive postmenopausal women with early-stage breast cancer. Clin Breast Cancer. 2007 Jun;7(8):608-18. doi: 10.3816/CBC.2007.n.018. PMID 17592673
- [Background] Buzdar A, Chlebowski R, Cuzick J, Duffy S, Forbes J, Jonat W, Ravdin P. Defining the role of aromatase inhibitors in the adjuvant endocrine treatment of early breast cancer. Curr Med Res Opin. 2006 Aug;22(8):1575-85. doi: 10.1185/030079906X120940. PMID 16870082
- [Background] Scott LJ, Keam SJ. Letrozole : in postmenopausal hormone-responsive early-stage breast cancer. Drugs. 2006;66(3):353-62. doi: 10.2165/00003495-200666030-00010. PMID 16526826
- [Background] Wardley AM. Emerging data on optimal adjuvant endocrine therapy: Breast International Group trial 1-98/MA.17. Clin Breast Cancer. 2006 Feb;6 Suppl 2:S45-50. doi: 10.3816/cbc.2006.s.003. PMID 16595026
- [Result] Leyland-Jones B, Gray KP, Abramovitz M, Bouzyk M, Young B, Long B, Kammler R, Dell'Orto P, Biasi MO, Thurlimann B, Harvey V, Neven P, Arnould L, Maibach R, Price KN, Coates AS, Goldhirsch A, Gelber RD, Pagani O, Viale G, Rae JM, Regan MM; BIG 1-98 Collaborative Group. ESR1 and ESR2 polymorphisms in the BIG 1-98 trial comparing adjuvant letrozole versus tamoxifen or their sequence for early breast cancer. Breast Cancer Res Treat. 2015 Dec;154(3):543-55. doi: 10.1007/s10549-015-3634-6. Epub 2015 Nov 21. PMID 26590813
- [Result] Colleoni M, Giobbie-Hurder A, Regan MM, Thurlimann B, Mouridsen H, Mauriac L, Forbes JF, Paridaens R, Lang I, Smith I, Chirgwin J, Pienkowski T, Wardley A, Price KN, Gelber RD, Coates AS, Goldhirsch A. Analyses adjusting for selective crossover show improved overall survival with adjuvant letrozole compared with tamoxifen in the BIG 1-98 study. J Clin Oncol. 2011 Mar 20;29(9):1117-24. doi: 10.1200/JCO.2010.31.6455. Epub 2011 Feb 14. PMID 21321298
- [Result] De Censi A, Sun Z, Thurlimann BJK, et al.: Bone mineral density (BMD) in participants (pts) of trial BIG 1-98 comparing adjuvant letrozole (L) versus tamoxifen (T) or their sequence. [Abstract] J Clin Oncol 29 (Suppl 15): A-516, 2011.
- [Result] Ejlertsen B, Aldridge J, Nielsen KV, Regan MM, Henriksen KL, Lykkesfeldt AE, Muller S, Gelber RD, Price KN, Rasmussen BB, Viale G, Mouridsen H; Danish Breast Cancer Cooperative Group the BIG 1-98 Collaborative Group and the International Breast Cancer Study Group. Prognostic and predictive role of ESR1 status for postmenopausal patients with endocrine-responsive early breast cancer in the Danish cohort of the BIG 1-98 trial. Ann Oncol. 2012 May;23(5):1138-1144. doi: 10.1093/annonc/mdr438. Epub 2011 Oct 10. PMID 21986093
- [Result] Huober JB, Cole BF, Wu J, et al.: Symptoms of endocrine treatment and outcome: A retrospective analysis of the monotherapy arms of the BIG 1-98 trial. [Abstract] J Clin Oncol 29 (Suppl 15): A-522, 2011.
- [Result] Phillips KA, Aldridge J, Ribi K, Sun Z, Thompson A, Harvey V, Thurlimann B, Cardoso F, Pagani O, Coates AS, Goldhirsch A, Price KN, Gelber RD, Bernhard J. Cognitive function in postmenopausal breast cancer patients one year after completing adjuvant endocrine therapy with letrozole and/or tamoxifen in the BIG 1-98 trial. Breast Cancer Res Treat. 2011 Feb;126(1):221-6. doi: 10.1007/s10549-010-1235-y. Epub 2010 Nov 3. PMID 21046229
- [Result] Regan MM, Neven P, Giobbie-Hurder A, Goldhirsch A, Ejlertsen B, Mauriac L, Forbes JF, Smith I, Lang I, Wardley A, Rabaglio M, Price KN, Gelber RD, Coates AS, Thurlimann B; BIG 1-98 Collaborative Group; International Breast Cancer Study Group (IBCSG). Assessment of letrozole and tamoxifen alone and in sequence for postmenopausal women with steroid hormone receptor-positive breast cancer: the BIG 1-98 randomised clinical trial at 8.1 years median follow-up. Lancet Oncol. 2011 Nov;12(12):1101-8. doi: 10.1016/S1470-2045(11)70270-4. Epub 2011 Oct 20. PMID 22018631
- [Result] Regan MM, Price KN, Giobbie-Hurder A, Thurlimann B, Gelber RD; International Breast Cancer Study Group and BIG 1-98 Collaborative Group. Interpreting Breast International Group (BIG) 1-98: a randomized, double-blind, phase III trial comparing letrozole and tamoxifen as adjuvant endocrine therapy for postmenopausal women with hormone receptor-positive, early breast cancer. Breast Cancer Res. 2011 May 26;13(3):209. doi: 10.1186/bcr2837. PMID 21635709
- [Result] Viale G, Regan MM, Dell'Orto P, Mastropasqua MG, Maiorano E, Rasmussen BB, MacGrogan G, Forbes JF, Paridaens RJ, Colleoni M, Lang I, Thurlimann B, Mouridsen H, Mauriac L, Gelber RD, Price KN, Goldhirsch A, Gusterson BA, Coates AS; BIG 1-98 Collaborative and International Breast Cancer Study Groups. Which patients benefit most from adjuvant aromatase inhibitors? Results using a composite measure of prognostic risk in the BIG 1-98 randomized trial. Ann Oncol. 2011 Oct;22(10):2201-7. doi: 10.1093/annonc/mdq738. Epub 2011 Feb 18. PMID 21335417
- [Result] Zaman K, Thurlimann B, Huober J, Schonenberger A, Pagani O, Luthi J, Simcock M, Giobbie-Hurder A, Berthod G, Genton C, Brauchli P, Aebi S; Swiss Group for Clinical Cancer Research (SAKK). Bone mineral density in breast cancer patients treated with adjuvant letrozole, tamoxifen, or sequences of letrozole and tamoxifen in the BIG 1-98 study (SAKK 21/07). Ann Oncol. 2012 Jun;23(6):1474-81. doi: 10.1093/annonc/mdr448. Epub 2011 Oct 14. PMID 22003243
- [Result] Antonov J, Popovici V, Delorenzi M, Wirapati P, Baltzer A, Oberli A, Thurlimann B, Giobbie-Hurder A, Viale G, Altermatt HJ, Aebi S, Jaggi R. Molecular risk assessment of BIG 1-98 participants by expression profiling using RNA from archival tissue. BMC Cancer. 2010 Feb 9;10:37. doi: 10.1186/1471-2407-10-37. PMID 20144231
- [Result] Phillips KA, Ribi K, Sun Z, Stephens A, Thompson A, Harvey V, Thurlimann B, Cardoso F, Pagani O, Coates AS, Goldhirsch A, Price KN, Gelber RD, Bernhard J. Cognitive function in postmenopausal women receiving adjuvant letrozole or tamoxifen for breast cancer in the BIG 1-98 randomized trial. Breast. 2010 Oct;19(5):388-95. doi: 10.1016/j.breast.2010.03.025. Epub 2010 Apr 10. PMID 20385495
- [Result] Ribi K, Aldridge J, Phillips K, et al.: Changes in cognitive function in postmenopausal women 1 year after completing adjuvant letrozole or tamoxifen in the Breast International Group (BIG) 1-98 trial. [Abstract] J Clin Oncol 28 (Suppl 15): A-527, 2010.
- [Result] BIG 1-98 Collaborative Group; Mouridsen H, Giobbie-Hurder A, Goldhirsch A, Thurlimann B, Paridaens R, Smith I, Mauriac L, Forbes J, Price KN, Regan MM, Gelber RD, Coates AS. Letrozole therapy alone or in sequence with tamoxifen in women with breast cancer. N Engl J Med. 2009 Aug 20;361(8):766-76. doi: 10.1056/NEJMoa0810818. PMID 19692688
- [Result] Giobbie-Hurder A, Price KN, Gelber RD; International Breast Cancer Study Group; BIG 1-98 Collaborative Group. Design, conduct, and analyses of Breast International Group (BIG) 1-98: a randomized, double-blind, phase-III study comparing letrozole and tamoxifen as adjuvant endocrine therapy for postmenopausal women with receptor-positive, early breast cancer. Clin Trials. 2009 Jun;6(3):272-87. doi: 10.1177/1740774509105380. PMID 19528136
- [Result] Rabaglio M, Sun Z, Price KN, Castiglione-Gertsch M, Hawle H, Thurlimann B, Mouridsen H, Campone M, Forbes JF, Paridaens RJ, Colleoni M, Pienkowski T, Nogaret JM, Lang I, Smith I, Gelber RD, Goldhirsch A, Coates AS; BIG 1-98 Collaborative and International Breast Cancer Study Groups. Bone fractures among postmenopausal patients with endocrine-responsive early breast cancer treated with 5 years of letrozole or tamoxifen in the BIG 1-98 trial. Ann Oncol. 2009 Sep;20(9):1489-1498. doi: 10.1093/annonc/mdp033. Epub 2009 May 27. PMID 19474112
- [Result] Regan MM, Colleoni M M, Giobbie-Hurder A, et al.: Adjusting for selective crossover in analyses of letrozole (Let) versus tamoxifen (Tam) in the BIG 1-98 trial. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-16, 2009.
- [Result] Ribi KE, Phillips KA, Sun Z, et al.: Cognitive function in postmenopausal women receiving adjuvant letrozole or tamoxifen in the Breast International Group (BIG) 1-98 trial. [Abstract] J Clin Oncol 27 (Suppl 15): A-510, 2009.
- [Result] Sun Z, Goldhirsch A, Price KN, Colleoni M, Ravaioli A, Simoncini E, Campbell I, Gelber RD, Towler M. Bone Quality Test (BQT) scores of fingernails in postmenopausal patients treated with adjuvant letrozole or tamoxifen for early breast cancer. Breast. 2009 Apr;18(2):84-8. doi: 10.1016/j.breast.2009.01.003. Epub 2009 Feb 24. PMID 19243946
- [Result] Viale G, Regan MM, Dell'Orto P, et al.: Central review of ER, PgR and HER2 in BIG 1-98 evaluating letrozole vs. letrozole followed by tamoxifen vs. tamoxifen followed by letrozole as adjuvant endocrine therapy for postmenopausal women with hormone receptor-positive breast cancer. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-76, 2009.
- [Result] Zaman K, Thürlimann B, Huober J, et al.: Modelling bone mineral density in Swiss breast cancer patients treated with letrozole, tamoxifen and sequences of letrozole and tamoxifen in the BIG 1-98 study (SAKK 21/07). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-5037, 2009.
- [Result] Crivellari D, Sun Z, Coates AS, Price KN, Thurlimann B, Mouridsen H, Mauriac L, Forbes JF, Paridaens RJ, Castiglione-Gertsch M, Gelber RD, Colleoni M, Lang I, Del Mastro L, Gladieff L, Rabaglio M, Smith IE, Chirgwin JH, Goldhirsch A. Letrozole compared with tamoxifen for elderly patients with endocrine-responsive early breast cancer: the BIG 1-98 trial. J Clin Oncol. 2008 Apr 20;26(12):1972-9. doi: 10.1200/JCO.2007.14.0459. Epub 2008 Mar 10. PMID 18332471
- [Result] Doughty JC. A review of the BIG results: the Breast International Group 1-98 trial analyses. Breast. 2008 Jan;17 Suppl 1:S9-S14. doi: 10.1016/S0960-9776(08)70003-1. PMID 18279765
- [Result] Mouridsen HT, Giobbie-Hurder A, Mauriac L, et al.: BIG 1-98: a randomized double-blind phase III study evaluating letrozole and tamoxifen given in sequence as adjuvant endocrine therapy for postmenopausal women with receptor-positive breast cancer. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-13, 2008.
- [Result] Rasmussen BB, Regan MM, Lykkesfeldt AE, Dell'Orto P, Del Curto B, Henriksen KL, Mastropasqua MG, Price KN, Mery E, Lacroix-Triki M, Braye S, Altermatt HJ, Gelber RD, Castiglione-Gertsch M, Goldhirsch A, Gusterson BA, Thurlimann B, Coates AS, Viale G; BIG 1-98 Collaborative and International Breast Cancer Study Groups. Adjuvant letrozole versus tamoxifen according to centrally-assessed ERBB2 status for postmenopausal women with endocrine-responsive early breast cancer: supplementary results from the BIG 1-98 randomised trial. Lancet Oncol. 2008 Jan;9(1):23-8. doi: 10.1016/S1470-2045(07)70386-8. Epub 2007 Dec 20. PMID 18083065
- [Result] Viale G, Giobbie-Hurder A, Regan MM, Coates AS, Mastropasqua MG, Dell'Orto P, Maiorano E, MacGrogan G, Braye SG, Ohlschlegel C, Neven P, Orosz Z, Olszewski WP, Knox F, Thurlimann B, Price KN, Castiglione-Gertsch M, Gelber RD, Gusterson BA, Goldhirsch A; Breast International Group Trial 1-98. Prognostic and predictive value of centrally reviewed Ki-67 labeling index in postmenopausal women with endocrine-responsive breast cancer: results from Breast International Group Trial 1-98 comparing adjuvant tamoxifen with letrozole. J Clin Oncol. 2008 Dec 1;26(34):5569-75. doi: 10.1200/JCO.2008.17.0829. Epub 2008 Nov 3. PMID 18981464
- [Result] Wardley AM. Understanding the BIG results: Insights from the BIG 1-98 trial analyses. Adv Ther. 2008 Dec;25(12):1257-75. doi: 10.1007/s12325-008-0128-5. PMID 19096768
- [Result] Coates AS, Keshaviah A, Thurlimann B, Mouridsen H, Mauriac L, Forbes JF, Paridaens R, Castiglione-Gertsch M, Gelber RD, Colleoni M, Lang I, Del Mastro L, Smith I, Chirgwin J, Nogaret JM, Pienkowski T, Wardley A, Jakobsen EH, Price KN, Goldhirsch A. Five years of letrozole compared with tamoxifen as initial adjuvant therapy for postmenopausal women with endocrine-responsive early breast cancer: update of study BIG 1-98. J Clin Oncol. 2007 Feb 10;25(5):486-92. doi: 10.1200/JCO.2006.08.8617. Epub 2007 Jan 2. PMID 17200148
- [Result] Mouridsen H, Keshaviah A, Coates AS, Rabaglio M, Castiglione-Gertsch M, Sun Z, Thurlimann B, Mauriac L, Forbes JF, Paridaens R, Gelber RD, Colleoni M, Smith I, Price KN, Goldhirsch A. Cardiovascular adverse events during adjuvant endocrine therapy for early breast cancer using letrozole or tamoxifen: safety analysis of BIG 1-98 trial. J Clin Oncol. 2007 Dec 20;25(36):5715-22. doi: 10.1200/JCO.2007.12.1665. Epub 2007 Nov 12. PMID 17998546
- [Result] Crivellari D, Sun Z, Coates AS, et al.: Aromatase inhibitors (AI) for elderly patients: efficacy, compliance and safety according to patient age in the BIG 1-98 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-9033, 501s, 2007.
- [Result] Koeberle D, Thuerlimann B. Letrozole as upfront endocrine therapy for postmenopausal women with hormone-sensitive breast cancer: BIG 1-98. Breast Cancer Res Treat. 2007;105 Suppl 1(Suppl 1):55-66. doi: 10.1007/s10549-007-9700-y. Epub 2007 Oct 3. PMID 17912636
- [Result] Mauriac L, Keshaviah A, Debled M, Mouridsen H, Forbes JF, Thurlimann B, Paridaens R, Monnier A, Lang I, Wardley A, Nogaret JM, Gelber RD, Castiglione-Gertsch M, Price KN, Coates AS, Smith I, Viale G, Rabaglio M, Zabaznyi N, Goldhirsch A; BIG 1-98 Collaborative Group; International Breast Cancer Study Group. Predictors of early relapse in postmenopausal women with hormone receptor-positive breast cancer in the BIG 1-98 trial. Ann Oncol. 2007 May;18(5):859-67. doi: 10.1093/annonc/mdm001. Epub 2007 Feb 14. PMID 17301074
- [Result] Monnier AM. The Breast International Group 1-98 trial: big results for women with hormone-sensitive early breast cancer. Expert Rev Anticancer Ther. 2007 May;7(5):627-34. doi: 10.1586/14737140.7.5.627. PMID 17492927
- [Result] Rasmussen BB, Regan MM, Lykkesfeldt AE, et al.: Central assessment of ER, PgR and HER2 in BIG 1-98 evaluating letrozole (L) compared to tamoxifen (T) as initial adjuvant endocrine therapy for postmenopausal women with hormone receptor-positive breast cancer. [Abstract] J Clin Oncol 25 (18 Suppl 20): A-538, 2007.
- [Result] Viale G, Regan MM, Maiorano E, Mastropasqua MG, Dell'Orto P, Rasmussen BB, Raffoul J, Neven P, Orosz Z, Braye S, Ohlschlegel C, Thurlimann B, Gelber RD, Castiglione-Gertsch M, Price KN, Goldhirsch A, Gusterson BA, Coates AS. Prognostic and predictive value of centrally reviewed expression of estrogen and progesterone receptors in a randomized trial comparing letrozole and tamoxifen adjuvant therapy for postmenopausal early breast cancer: BIG 1-98. J Clin Oncol. 2007 Sep 1;25(25):3846-52. doi: 10.1200/JCO.2007.11.9453. Epub 2007 Aug 6. PMID 17679725
- [Result] Forbes JF. The use of early adjuvant aromatase inhibitor therapy: contributions from the BIG 1-98 letrozole trial. Semin Oncol. 2006 Apr;33(2 Suppl 7):S2-7. doi: 10.1053/j.seminoncol.2006.03.026. PMID 16730270
- [Result] Breast International Group (BIG) 1-98 Collaborative Group; Thurlimann B, Keshaviah A, Coates AS, Mouridsen H, Mauriac L, Forbes JF, Paridaens R, Castiglione-Gertsch M, Gelber RD, Rabaglio M, Smith I, Wardley A, Price KN, Goldhirsch A. A comparison of letrozole and tamoxifen in postmenopausal women with early breast cancer. N Engl J Med. 2005 Dec 29;353(26):2747-57. doi: 10.1056/NEJMoa052258. PMID 16382061
- [Derived] Gregg JR, Zhang X, Chapin BF, Ward JF, Kim J, Davis JW, Daniel CR. Adherence to the Mediterranean diet and grade group progression in localized prostate cancer: An active surveillance cohort. Cancer. 2021 Mar 1;127(5):720-728. doi: 10.1002/cncr.33182. Epub 2021 Jan 7. PMID 33411364
- [Derived] Leone JP, Cole BF, Regan MM, Thurlimann B, Coates AS, Rabaglio M, Giobbie-Hurder A, Gelber RD, Ejlertsen B, Harvey VJ, Neven P, Lang I, Bonnefoi H, Wardley A, Goldhirsch A, Di Leo A, Colleoni M, Vaz-Luis I, Lin NU. Clinical behavior of recurrent hormone receptor-positive breast cancer by adjuvant endocrine therapy within the Breast International Group 1-98 clinical trial. Cancer. 2021 Mar 1;127(5):700-708. doi: 10.1002/cncr.33318. Epub 2020 Dec 8. PMID 33290610
- [Derived] Luen SJ, Asher R, Lee CK, Savas P, Kammler R, Dell'Orto P, Biasi OM, Demanse D, Hackl W, Thuerlimann B, Viale G, Di Leo A, Colleoni M, Regan MM, Loi S. Identifying oncogenic drivers associated with increased risk of late distant recurrence in postmenopausal, estrogen receptor-positive, HER2-negative early breast cancer: results from the BIG 1-98 study. Ann Oncol. 2020 Oct;31(10):1359-1365. doi: 10.1016/j.annonc.2020.06.024. Epub 2020 Jul 8. PMID 32652112
- [Derived] Kensler KH, Regan MM, Heng YJ, Baker GM, Pyle ME, Schnitt SJ, Hazra A, Kammler R, Thurlimann B, Colleoni M, Viale G, Brown M, Tamimi RM. Prognostic and predictive value of androgen receptor expression in postmenopausal women with estrogen receptor-positive breast cancer: results from the Breast International Group Trial 1-98. Breast Cancer Res. 2019 Feb 22;21(1):30. doi: 10.1186/s13058-019-1118-z. PMID 30795773
- [Derived] Ruhstaller T, Giobbie-Hurder A, Colleoni M, Jensen MB, Ejlertsen B, de Azambuja E, Neven P, Lang I, Jakobsen EH, Gladieff L, Bonnefoi H, Harvey VJ, Spazzapan S, Tondini C, Del Mastro L, Veyret C, Simoncini E, Gianni L, Rochlitz C, Kralidis E, Zaman K, Jassem J, Piccart-Gebhart M, Di Leo A, Gelber RD, Coates AS, Goldhirsch A, Thurlimann B, Regan MM; members of the BIG 1-98 Collaborative Group and the International Breast Cancer Study Group. Adjuvant Letrozole and Tamoxifen Alone or Sequentially for Postmenopausal Women With Hormone Receptor-Positive Breast Cancer: Long-Term Follow-Up of the BIG 1-98 Trial. J Clin Oncol. 2019 Jan 10;37(2):105-114. doi: 10.1200/JCO.18.00440. Epub 2018 Nov 26. PMID 30475668
- [Derived] Luen SJ, Asher R, Lee CK, Savas P, Kammler R, Dell'Orto P, Biasi OM, Demanse D, JeBailey L, Dolan S, Hackl W, Thuerlimann B, Viale G, Colleoni M, Regan MM, Loi S. Association of Somatic Driver Alterations With Prognosis in Postmenopausal, Hormone Receptor-Positive, HER2-Negative Early Breast Cancer: A Secondary Analysis of the BIG 1-98 Randomized Clinical Trial. JAMA Oncol. 2018 Oct 1;4(10):1335-1343. doi: 10.1001/jamaoncol.2018.1778. PMID 29902286
- [Derived] Dowsett M, Sestak I, Regan MM, Dodson A, Viale G, Thurlimann B, Colleoni M, Cuzick J. Integration of Clinical Variables for the Prediction of Late Distant Recurrence in Patients With Estrogen Receptor-Positive Breast Cancer Treated With 5 Years of Endocrine Therapy: CTS5. J Clin Oncol. 2018 Jul 1;36(19):1941-1948. doi: 10.1200/JCO.2017.76.4258. Epub 2018 Apr 20. PMID 29676944
- [Derived] Chirgwin JH, Giobbie-Hurder A, Coates AS, Price KN, Ejlertsen B, Debled M, Gelber RD, Goldhirsch A, Smith I, Rabaglio M, Forbes JF, Neven P, Lang I, Colleoni M, Thurlimann B. Treatment Adherence and Its Impact on Disease-Free Survival in the Breast International Group 1-98 Trial of Tamoxifen and Letrozole, Alone and in Sequence. J Clin Oncol. 2016 Jul 20;34(21):2452-9. doi: 10.1200/JCO.2015.63.8619. Epub 2016 May 23. PMID 27217455
- [Derived] Ignatiadis M, Azim HA Jr, Desmedt C, Veys I, Larsimont D, Salgado R, Lyng MB, Viale G, Leyland-Jones B, Giobbie-Hurder A, Kammler R, Dell'Orto P, Rothe F, Laios I, Ditzel HJ, Regan MM, Piccart M, Michiels S, Sotiriou C. The Genomic Grade Assay Compared With Ki67 to Determine Risk of Distant Breast Cancer Recurrence. JAMA Oncol. 2016 Feb;2(2):217-24. doi: 10.1001/jamaoncol.2015.4377. PMID 26633571
- [Derived] Munzone E, Giobbie-Hurder A, Gusterson BA, Mallon E, Viale G, Thurlimann B, Ejlertsen B, MacGrogan G, Bibeau F, Lelkaitis G, Price KN, Gelber RD, Coates AS, Goldhirsch A, Colleoni M; International Breast Cancer Study Group and the BIG 1-98 Collaborative Group. Outcomes of special histotypes of breast cancer after adjuvant endocrine therapy with letrozole or tamoxifen in the monotherapy cohort of the BIG 1-98 trial. Ann Oncol. 2015 Dec;26(12):2442-9. doi: 10.1093/annonc/mdv391. Epub 2015 Sep 19. PMID 26387144
- [Derived] Metzger Filho O, Giobbie-Hurder A, Mallon E, Gusterson B, Viale G, Winer EP, Thurlimann B, Gelber RD, Colleoni M, Ejlertsen B, Debled M, Price KN, Regan MM, Coates AS, Goldhirsch A. Relative Effectiveness of Letrozole Compared With Tamoxifen for Patients With Lobular Carcinoma in the BIG 1-98 Trial. J Clin Oncol. 2015 Sep 1;33(25):2772-9. doi: 10.1200/JCO.2015.60.8133. Epub 2015 Jul 27. PMID 26215945
- [Derived] Leyland-Jones B, Gray KP, Abramovitz M, Bouzyk M, Young B, Long B, Kammler R, Dell'Orto P, Biasi MO, Thurlimann B, Lyng MB, Ditzel HJ, Harvey VJ, Neven P, Treilleux I, Rasmussen BB, Maibach R, Price KN, Coates AS, Goldhirsch A, Pagani O, Viale G, Rae JM, Regan MM. CYP19A1 polymorphisms and clinical outcomes in postmenopausal women with hormone receptor-positive breast cancer in the BIG 1-98 trial. Breast Cancer Res Treat. 2015 Jun;151(2):373-84. doi: 10.1007/s10549-015-3378-3. Epub 2015 May 3. PMID 25935582
- [Derived] Huober J, Cole BF, Rabaglio M, Giobbie-Hurder A, Wu J, Ejlertsen B, Bonnefoi H, Forbes JF, Neven P, Lang I, Smith I, Wardley A, Price KN, Goldhirsch A, Coates AS, Colleoni M, Gelber RD, Thurlimann B; BIG 1-98 Collaborative and International Breast Cancer Study Groups. Symptoms of endocrine treatment and outcome in the BIG 1-98 study. Breast Cancer Res Treat. 2014 Jan;143(1):159-69. doi: 10.1007/s10549-013-2792-7. Epub 2013 Dec 5. PMID 24305979
- [Derived] Regan MM, Leyland-Jones B, Bouzyk M, Pagani O, Tang W, Kammler R, Dell'orto P, Biasi MO, Thurlimann B, Lyng MB, Ditzel HJ, Neven P, Debled M, Maibach R, Price KN, Gelber RD, Coates AS, Goldhirsch A, Rae JM, Viale G; Breast International Group (BIG) 1-98 Collaborative Group. CYP2D6 genotype and tamoxifen response in postmenopausal women with endocrine-responsive breast cancer: the breast international group 1-98 trial. J Natl Cancer Inst. 2012 Mar 21;104(6):441-51. doi: 10.1093/jnci/djs125. Epub 2012 Mar 6. PMID 22395644
- [Derived] Chirgwin J, Sun Z, Smith I, Price KN, Thurlimann B, Ejlertsen B, Bonnefoi H, Regan MM, Goldhirsch A, Coates AS; BIG 1-98 Collaborative and International Breast Cancer Study Groups. The advantage of letrozole over tamoxifen in the BIG 1-98 trial is consistent in younger postmenopausal women and in those with chemotherapy-induced menopause. Breast Cancer Res Treat. 2012 Jan;131(1):295-306. doi: 10.1007/s10549-011-1741-6. Epub 2011 Sep 4. PMID 21892704